CLINICAL TRIAL: NCT00488761
Title: A Multicenter, Open Label Study to Evaluate the Safety and Efficacy of Tigecycline to Treat Complicated Skin and Skin Structure Infections (cSSSI) in Hospitalized Patients
Brief Title: Study Evaluating the Safety and Efficacy of Tigecycline in Hospitalized Patients With cSSSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101993
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Skin Diseases, Infectious
Keywords: Tigecycline; cSSSI; complicated skin and skin structure infections
MeSH Terms: conditions — Skin Diseases, Infectious | interventions — Tigecycline

INTERVENTIONS:
Drug: Tigecycline

SUMMARY:
Tigecycline's activity against resistant organisms, as well as significant coverage of both gram-positive and gram-negative bacteria, may provide a valuable therapeutic alternative in treating patients with complicated skin and/or skin structure infections.

DETAILED DESCRIPTION:
To evaluate the safety and the efficacy of tigecycline in treating hospitalized patients with complicated skin and/or skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized male and female patients, 18 years of age or older.
* Anticipated need for intravenous antibiotic therapy of 5 days or longer.
* Patients known or suspected to have a complicated skin and skin structure infection.

Exclusion Criteria:

* Patients with any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy could be completed.
* Patients with severely impaired arterial blood supply and insufficiency such that the likelihood of amputation of the infected anatomical site within one month is likely.
* Infected diabetic foot ulcers or decubitus ulcers where the infection is present for greater than one week's duration or chronically infected decubitus ulcers in patients who can not be compliant with measures necessary for chronic wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the clinical response for all clinically evaluable patients (primary population) at the test-of-cure visit

SECONDARY OUTCOMES:
microbiological response at the patient level microbiological response at the pathogen level clinical cure rates by baseline pathogen response rates for patients with polymicrobial and monomicrobial infections

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Taiwan, medinfo@wyeth.com
Locations (1):
- Multiple Cities, Taiwan